CLINICAL TRIAL: NCT05671445
Title: An Open, Multineutral Study Evaluating the Safety and Efficacy of CM326 in the Long-term Treatment of Adult Subjects With Atopic Dermatitis
Brief Title: The Study of CM326 in Adult Subjects With Atopic Dermatitis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Keymed Biosciences Co.Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CM326-101105
Record Dates: First submitted 2022-12-26; First posted 2023-01-04 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-03

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CM326 (Experimental): CM326 injection, subcutaneous (SC)
  Interventions: Biological: CM326

INTERVENTIONS:
Biological: CM326 — CM326 injection

SUMMARY:
This is a open-label, multi-center study to evaluate the safety and efficacy of CM326 in atopic adrmatitis subjects.

DETAILED DESCRIPTION:
The study consists of 3 periods, a up-to-4-week Screening Period, a 52-week Treatment Period and a 8-week Safety Follow-up Period.

ELIGIBILITY:
Inclusion Criteria:

* With confirmed Atopic Dermatitis (AD) at the screening.
* Have the ability to understand the nature of the study and voluntarily sign the informed consent.
* Be able to communicate well with investigators and follow up protocol requirements.
* The subjects agreed to use highly effective contraceptive measures during the study.

Exclusion Criteria:

* Not enough washing-out period for previous therapy.
* Received allergen specific immunotherapy (desensitization) within 6 months prior to baseline.
* Major surgery is planned during the study period.
* Women who are pregnant or breastfeeding, or who plan to become pregnant during the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-02-09 (Actual); Primary Completion 2024-03-28 (Estimated); Study Completion 2025-03-28 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events | at week 52
  Incidence of treatment-emergent Adverse events related to CM326

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University People's hospital, Beijing, China